# The Effect of Dipeptidyl Peptidase IV Inhibition on Growth Hormone-Mediated Vasodilation

Jessica K. Devin, MD MSCI



# **Table of Contents:**

- 1.0 Background and Previous Human Studies
- 2.0 Rationale and Specific Aims
- 3.0 Inclusion/Exclusion Criteria
- 4.0 Enrollment/Randomization
- **5.0 Study Procedures**
- 6.0 Risks
- 7.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others
- 8.0 Study Withdrawal/Discontinuation
- 9.0 Statistical Considerations
- **10.0** Privacy/Confidentiality Issues
- 11.0 Follow-up and Record Retention

## 1. Background and Previous Human Studies

Dipeptidyl peptidase IV (DPPIV) is a ubiquitously expressed cell surface serine protease which cleaves a dipeptide from the N-terminus of its polypeptide substrates containing a proline or alanine at the second residue. Interest in this peptidase and its pharmacological inhibition has arisen due to its proteolytic inactivation of the incretin hormones and the role this plays in glucose homeostasis. Selective DPPIV inhibitors improve glycemic control in patients with type 2 diabetes mellitus by decreasing the degradation of the incretin hormones glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP).(1;2) The DPPIV inhibitor sitagliptin was approved by the FDA in 2006 as a once daily oral medication to lower blood sugar levels in patients with type 2 diabetes mellitus. Two additional DPPIV inhibitors have since received FDA approval: saxagliptin (2009) and linagliptin (2011). The direct and indirect effects of these inhibitors on cardiovascular function remain an active area of investigation.

GLP-1 also promotes endothelium-dependent vasodilation in the human vasculature in subjects with type 2 diabetes and stable coronary artery disease. In addition to preventing the degradation of the incretin hormones, DPPIV inhibitors prevent the degradation of other peptides with a penultimate proline or alanine including but not limited to the vasodilators substance P as well as BNP and the neurotransmitter neuropeptide Y.(3;4) Our group has previously demonstrated that five day treatment with sitagliptin significantly decreased mean arterial pressure in subjects with metabolic syndrome.(5) Others have reported that acute sitagliptin treatment reduces 24 hour ambulatory blood pressure in non-diabetic patients with mild to moderate hypertension.(6) It has recently been demonstrated in an animal model and *in vitro* that acute DPPIV inhibition leads to vascular relaxation via a GLP-1 independent mechanism involving nitric oxide release mediated by Akt dependent phosphorylation of endothelial nitric oxide synthase.(7)

DPPIV inhibitors could affect blood pressure and vascular function in part by their effect on the somatotropic axis. Pituitary growth hormone releasing hormone (GHRH), also known as growth hormone-releasing factor (GRF) is a substrate of DPPIV, which rapidly cleaves GRF(1-44)-NH<sub>2</sub> to the biologically inactive GRF (3-44)-NH<sub>2</sub> at Ala<sup>2</sup>-Asp<sup>3</sup>.(1;2) Conversion to GRF (3-44)-NH<sub>2</sub> is blocked *in vitro* by diprotin A, a DPPIV competitive inhibitor.(8) Human GRF is produced in the hypothalamus and stimulates the release of the growth hormone (GH) from somatotrope cells within the anterior pituitary gland; the active portion of the molecule resides in the first 29 amino acid residues. Opposing the actions of GRF, the hypothalamic hormone somatostatin inhibits the release of GRF.(9) Growth hormone circulates throughout the body exerting its

numerous effects both directly and indirectly via the hepatic production of insulin-like growth factor-1 (IGF-1). DPPIV proteolysis plays a major role in the degradation and inactivation of human GRF *in vivo*.(2) Thus, we hypothesize that inhibition of DPPIV will result in decreased GRF degradation and augmentation of the somatotropic axis *in vivo* in humans.

The direct vascular effects of GH and its downstream mediator IGF-1 are wellestablished. Systemic and arterial GH infusion increases forearm blood flow in healthy subjects independent of systemic and local IGF-1 production.(10;11) This vasodilation is reversed by infusion of the nitric oxide inhibitor, L-N-monomethylarginine (L-NMMA).(10) Furthermore, growth hormone receptors are present in abundance on human endothelial cells. Incubation of endothelial cells with GH in vitro increases the phosphorylation and activity of endothelial nitric oxide synthase (eNOS) resulting in increased formation of nitric oxide (NO). NO is formed by endothelial nitric oxide synthase (eNOS) within the endothelial cells of the vasculature and then diffuses to underlying smooth muscle cells where it increases vasodilation via cGMP production and decreases inflammation and platelet aggregation.(12-14) Growth hormone treatment also contributes to vascular integrity by enhancing NO-mediated mobilization of endothelial progenitor cells in healthy individuals.(15;16) The exact mechanism(s) through which GH regulates eNOS remain unclear. Evidence exists for both an IGF-1 mediated activation of eNOS involving the serine/threonine Akt phosphorylationdependent kinase as well as a direct GH-mediated activation of both Akt and JAK-STAT (Janus kinase-signal transducer and activator of transcription) pathways.(17)

Interestingly, individuals with hypopituitarism experience increased cardiovascular and cerebrovascular morbidity and mortality as well as an increased prevalence of cardiovascular risk factors, despite adequate steroid and thyroid hormone replacement though lacking in growth hormone replacement.(18-20) The PI has demonstrated that adults with growth hormone deficiency also demonstrate alterations in plasma fibrinolytic balance, as compared to gender, age, and body mass index-matched controls.(21) Several prospective studies in adults with hypopituitarism have demonstrated that GH replacement improves cardiac function, intima-media thickness, endothelial function, and vascular reactivity as well as various biochemical markers of cardiovascular and metabolic disease including fat distribution and inflammatory cytokines.(22-27) Furthermore, GH deficient adults exhibit low levels of metabolites of systemic NO production; and GH replacement therapy normalizes biomarkers of NO.(16;28;29) Many of the adverse cardiovascular factors observed in GH deficient individuals are accordingly attributed to inadequate vascular NO bioavailability which can be reversed with GH treatment.

Patients with the cardiovascular risk factors of hypertension, hyperlipidemia, diabetes mellitus or tobacco use demonstrate endothelial dysfunction characterized by the inability of the endothelium to generate adequate amounts of NO.(14) Basal NO-mediated dilatation in the forearm arterial bed of patients with insulin-dependent diabetes is impaired as assessed by venous occlusion plethysmography.(30) The impairment in endothelial function in experimental animals and humans with diabetes mellitus is attributed to reduced NOS activity and/or NO availability as well as the accompanying increased production of reactive oxygen species. This characteristic endothelial dysfunction has been implicated in the pathogenesis of diabetic vascular disease.(31)

This aim promises to provide important new data regarding how DPPIV inhibition affects the somatotropic axis in healthy adults. Given the known effects that growth hormone and IGF-1 have on endothelial function as well as cardiovascular and metabolic markers, an augmentation of this axis may positively impact vascular function in the diabetic population. None of our currently available anti-glycemic agents offer this benefit. Data from the Framingham Heart Study demonstrates a negative correlation between circulating IGF-1 and insulin resistance in a community based sample.(32) GRF-induced GH secretion is blunted in premenopausal women with hyperlipidemia and insulin resistance.(33) Thus derangements in the somatotropic axis have previously been described in individuals at risk for the development of diabetes.

Adults with diabetes demonstrate heart disease death rates two to four times higher than adults without diabetes ("Diabetes Statistics" American Diabetes Association; www.diabetes.org); thus DPPIV inhibitors may potentially represent a novel therapy that is simultaneously able to confer both a glycemic and vascular benefit in this at-risk population. We therefore expect that findings from this study will lead to further investigations regarding currently unrecognized but significant vascular effects of this relatively new class of medications increasingly used in the diabetic population.

### 2. Rationale and Specific Aims

This study tests the hypothesis that DPPIV inhibition will favorably augment the somatotropic axis in healthy individuals by decreasing the degradation of GRF by DPPIV. This study specifically establishes the effect of acute DPP4 inhibition on arginine-stimulated GH secretion and GH-mediated blood flow in healthy humans. Arginine decreases inhibitory hypothalamic somatostatin secretion, allowing the primary stimulus of GH secretion to be GHRH. We will study healthy adults to obtain maximal GH signal in this proof-of-concept initial aim, given that obesity diminishes the GH response to pharmacologic stimuli.

- -Aim 1A tests the hypothesis that acute DPP4 inhibition will increase stimulated GH secretion in healthy lean adults by decreasing the degradation of GHRH.
- -Aim 1B tests the hypothesis that decreased degradation of GHRH during acute DPP4 inhibition will result in an increase in endothelium-dependent vasodilation mediated by GH, and independent from GLP-1.

This study promises to provide novel data regarding how this increasingly used class of anti-diabetic drugs could modulate vascular function. Given the known changes within the somatotropic axis in the setting of insulin resistance, further studies may wish to evaluate the effect of DPPIV inhibition in individuals with the metabolic syndrome.



### 3. Inclusion/Exclusion Criteria

Forty-two (fourteen per group) healthy, non-smoking subjects (31 females and 11 males), age 18 through 40 years of age will participate in this randomized, double-blind, placebo-controlled crossover study. Subjects taking medications other than multivitamins will be excluded. Pregnancy will be excluded in women of child-bearing age by serum β-HCG.

### **Inclusion Criteria**

- Age 18 to 40 years inclusive
- BMI  $\leq$  25 kg/m<sup>2</sup>
- For female subjects:
  - o Status-post surgical sterilization, or
  - $_{\odot}$  If of child-bearing potential, utilization of a barrier method of birth control following negative serum  $\beta$ -HCG at screening visit and on every study day

### **Exclusion Criteria**

- Smoking
- Type 1 or Type 2 Diabetes Mellitus, as defined by a fasting glucose of 126 mg/dL or greater at the time of screening visit or the use of anti-diabetic medication
- Hypertension, as defined by an untreated seated SBP greater than 140 mmHg and/or an untreated DBP greater than 90 mmHg at the time of screening visit or the use of anti-hypertensive medication
- History of reported or recorded hypoglycemia (plasma glucose < 70 mg/dL)</li>
- Pregnancy and/or Breast-Feeding
- Use of any medication other than multivitamin, including use of transdermal as well as oral hormone replacement therapy
- Anemia defined as hematocrit <35% at screening visit</li>
- Cardiovascular or cerebrovascular disease, including history of myocardial infarction, history of congestive heart failure, history of stroke
- Pulmonary Hypertension
- Abnormal thyroid hormone levels (TSH) at the time of screening visit
- Abnormal serum IGF-1 at the time of screening visit
- Impaired renal function, defined as eGFR <60 mL/min/1.73M<sup>2</sup>
- Impaired hepatic function (AST or ALT > 2 X upper limit of normal range)
- Treatment with an investigational drug in the 1 month preceding the study

### 4. Enrollment/Randomization

Subjects will be randomly assigned to treatment order (**see below table**) for each pair of visits using a block randomization algorithm with a block size of 2. study biostatistician, will provide an allocation schedule. The Vanderbilt Investigational Drug Service will be responsible for the storage, preparation, and labeling of all

investigational agents and for maintaining accurate drug storage and dispending logs. A Clinical Research Pharmacist in the Vanderbilt Investigational Drug Service will devise standard operating procedures for the pharmacy to follow with regard to preparing, labeling, blinding, and dispensing study drug. The Investigational Drug Service will retain a secure set of sealed envelopes containing the treatment assignment.

Randomized subjects who do not complete the whole protocol for any reason will be replaced.

| Aim 1A<br>Randomization | Anticipated<br>Result | Aim 1B Randomization | Anticipated Result |
|---|---|---|---|
| | | Group A (N=14) Sitagliptin + [L-NMMA vs. Placebo] | Endothelium-dependent<br>vasodilation mediated by<br>Arginine, GH, and GLP-1<br>blocked |
| Sitagliptin vs. Placebo (N=42) | Sitagliptin increases stimulated GH secretion and FBF | Group B (N=14) Sitagliptin + [GH Receptor Antagonist vs. Placebo] | GH mediated vasodilation blocked |
| | | Group C (N=14) Sitagliptin + [GLP-1 Receptor Antagonist vs. Placebo] | Endothelium-dependent and independent vasodilation mediated by GLP-1 blocked |

# 5. Study Procedures



Aim 1 A Study Protocol
(Two study days separated by a 2 week washout)

The figure above illustrates the **Aim 1A** study protocol for **Groups A** and **C** (Group B has completed Aim 1A). Each subject will undergo two study days separated by at least a 2 week wash-out. Seventy-two hours prior to each study day, subjects will start once daily study drug (sitagliptin 100 mg by mouth or matching placebo), following a negative pregnancy test obtained in the Vanderbilt Clinical Research Center (CRC), as applicable. This duration and dose of sitagliptin was chosen to achieve steady-state with significant inhibition of DPP4 activity.(34) On each day, subjects will report to the Vanderbilt Clinical Research Center (CRC) in the morning after an overnight fast and having abstained from exercise that morning. Subjects will be studied in the supine position in a temperature-controlled room. All subjects will receive a peripheral venous

catheter in the non-dominant arm for infusion of arginine as well as a peripheral venous catheter in the contra-lateral arm for repeated blood sampling. Normal saline will be infused into the catheter in the non-dominant arm prior to arginine administration for purposes of keeping the vein open. Subjects will then be given their 4<sup>th</sup> dose of study drug. One hour after administration of study drug we will measure baseline forearm blood flow (FBF, see below) and obtain baseline venous blood samples (see below). We will infuse arginine (30 grams) intravenously over 30 minutes. We have chosen this dose of arginine, previously used in the clinical setting to diagnose GH deficiency, to yield a peak plasma GH level of 10 ng/mL 30minutes after completion of arginine infusion.(35;36). Immediately following arginine administration we will repeat measurements of forearm blood flow every 30 minutes and venous blood sampling every 15 minutes up to 150 minutes after arginine infusion. The protocol will be repeated following a 2-week washout using the opposite study drug (sitagliptin or matching placebo). Both blood pressure and heart rate will be continuously monitored throughout each study day. At the completion of each study day subjects will be fed lunch prior to discharge from the CRC.



\*\*Antagonists include L-NMMA (Group A), GH Receptor Blocker (Group B), GLP-1 Receptor Blocker (Group C)

The figure above illustrates *Aim 1B.* If an effect of sitagliptin on FBF is observed, subjects will be invited to return for 2 additional study visits (Study Visits 3 and 4) in order to elucidate the mechanism underlying the increase in FBF. Study Visit 3 will occur at least 8 weeks after Study Visit 2. Subjects will be given DPP4 inhibitor as well as double-blinded antagonist vs. placebo (*see previous table*) on each study days. In **Group B**, DPP4 inhibition will be given as a single oral dose (sitagliptin 200 mg) on each study day; a minimum of 4 weeks will separate study days. In **Groups A and C**, DPP4 inhibition will be given as 100 mg sitagliptin by mouth daily, starting 72 hours prior to each study day with the 4<sup>th</sup> dose given on the study day; a minimum two-week washout will separate study days. Venous sampling will occur following assessment of forearm blood flow. All other study procedures will take place as previously described. Details regarding the dose and administration of each antagonist are provided below.

### Forearm Blood Flow Measurements

FBF will be measured using mercury-in-silastic strain-gauge plethysmography. The wrist is supported in a sling to raise the level of the forearm to above the level of the

atrium, and a strain gauge is placed in the widest part of the forearm. The strain gauge is connected to a plethysmograph (model EC-4, D.E. Hokanson, Issaquah, WA), calibrated to measure the percent change in volume and connected to a chart recorder to record flow measurements. For each measurement, a cuff placed around the upper arm is inflated to 40 mmHg with a rapid cuff inflator (model E-10, Hokanson) to occlude venous outflow from the extremity. The hand is excluded from the measurement of blood flow by inflation of a pediatric sphygmomanometer cuff to 200 mmHg around the wrist during measurement of FBF. Flow measurements are recorded for approximately 7 secs/15 secs, and the slope is derived from the first 3-4 pulses; 7 readings are obtained for each mean.

### Venous Blood Sampling

Following measurement of FBF, venous samples will be obtained prior to arginine administration and immediately as the completion of arginine 30 minute infusion. Venous samples will then be obtained every 15 minutes up to 150 minutes following completion of arginine infusion in Aim 1A. In Aim 1B, venous samples will be obtained before and following arginine infusion at 8 designated timepoints. Samples may be analyzed for ADMA, arginine, GH, insulin, glucose, GLP-1, DPP4 activity and antigen, cGMP, PAI-1 antigen, tPA activity and IGF-1.

The dose of GH receptor antagonist (pegvisomant 80 mg given subcutaneously 72 hours prior to each study day in Aim 1B) was chosen as 80 mg of pegvisomant produces maximal drug levels 72 hours following administration and a reduction in free IGF-1 comparable to that observed in GH deficiency, thus indicative of efficient GH receptor blockade and a state of acute GH deficiency.(37;38) Pegvisomant is a GH analog that disables signal transduction through the GH receptor and thereby functions as a receptor antagonist. This selective blockade allows us to examine the effects of GH secretion in the absence of cofounders such as changes in IGF-1 secretion and body composition which may accompany chronic GH deficiency. This method of achieving acute GH blockade has been reported to safely and effectively study GH secretion in a variety of metabolic conditions and to evaluate the effect of GH secretion on cardiovascular risk markers.(37-39)

The dose of GLP-1 receptor antagonist (Exendin-(9-39) IV bolus of 7500 pmol/kg over 1 minute at time 0 (Aim 1B) followed by continuous infusion of 750 pmol/kg/min for 150 minutes) was chosen as this dose elicits blockade of GLP-1 action at its receptor in healthy volunteers during a fixed blood glucose, as measured by augmented post-prandial glucagon secretion, a blunted increase in post-prandial insulin secretion, and a significant increase in post-prandial GLP-1 secretion.(40-

42)The timing of Exendin-(9-39) infusion may be adjusted pending results of Aim1A to coincide with the timing of peak FBF response.

The dose and timing of the nitric oxide synthase inhibitor, L-NMMA (3mg/kg priming IV infusion over 15 minutes given prior to Arginine infusion in Aim 1B and then continued at 6 mg/kg over an additional 120 minutes) has been selected to achieve peak hemodynamic response 15 minutes after priming dose and maintain hemodynamic effects for up to one hour after completion of infusion.(43;44) Doses up to 13.5 mg/kg IV have safely been given to healthy adults. (44-46) The elimination half-life of L-NMMA is approximately 60 minutes.(43) Co-infusion of a total dose of 6.5 mg/kg L-NMMA with L-arginine has not been shown to influence L-arginine-stimulated GH secretion.(47)

### 6. Risks

- 1. Repeated blood sampling from venous catheters may cause bleeding or infection.
- 2. Frequent blood draws can cause anemia.
- 3. Insertion of venous catheters may cause bleeding, bruising, or infection.
- 4. Arginine has previously been used to diagnose growth hormone deficiency (IV, 30 grams).(36) After completion of infusion, L-arginine plasma concentration rapidly decreases within 30 minutes to 47% of the maximum level. (43) Possible side effects include flushing, nausea and vomiting, headache, numbness and local venous irritation. Rarely, a burn-like reaction or injury to the skin requiring surgery has been reported. Rarely, allergic reaction has been reported.
- 5. Sitagliptin Drugs like sitagliptin can cause lowered blood sugar (common) in individuals with high blood sugar (diabetes). This can result in dizziness, nausea, shaking, sweating, fast heartbeat, vision changes, headache, anxiety, tiredness, or confusion. It can rarely cause fainting, seizures, or coma. Other side effects are pancreatitis (damage to the pancreas), kidney damage (which can be life threatening), allergic reaction (which can be life threatening), rash, and liver damage (which can be life threatening). The FDA is warning that dipeptidyl peptidase-4 (DPP-4) inhibitors such as sitagliptin, saxagliptin, linagliptin, and alogliptin may cause joint pain that can be severe and

disabling. After the patients discontinued the DPP-4 inhibitor medicine, their symptoms were relieved, usually in less than a month. Some patients developed severe joint pain again when they restarted the same medicine or another DPP-4 inhibitor.

- 6. The dose of GH receptor antagonist (Pegvisomant 80 mg given subcutaneously 72 hours prior to each study day in Aim 1B, Group B only) was chosen as 80 mg of pegvisomant produces maximal drug levels 72 hours following administration and a reduction in free IGF-1 comparable to that observed in GH deficiency, thus indicative of efficient GH receptor blockade and a state of acute GH deficiency.(37;38) Pegvisomant is a GH analog that disables signal transduction through the GH receptor and thereby functions as a receptor antagonist. This selective blockade allows us to examine the effects of GH secretion in the absence of cofounders such as changes in IGF-1 secretion and body composition which may accompany chronic GH deficiency. This method of achieving acute GH blockade has been reported to safely and effectively study GH secretion in a variety of metabolic conditions and to evaluate the effect of GH secretion on cardiovascular risk markers.(37-39) Side effects in patients taking this medication on a daily basis may include pain and reaction at the injection site, flu-like symptoms, nausea, and diarrhea (common). Rarely, swelling, dizziness, sinusitis and elevations in liver tests have been reported with repeated use.
- 7. Exendin-(9-39) (IND \_\_\_\_\_)-is an investigational agent (Clinalfa®, Bachem Distribution Services; Weil am Rhein, Germany) that will be infused intravenously following dissolution in 0.25% human serum albumin. Salehi et. al. have not experienced any untoward effects with the use of this antagonist in healthy participants, those with Type 2 diabetes mellitus, or history of gastric bypass.(40;42;48) Deane et. al. reported that blockade of GLP-1 action was associated with accelerated gastric emptying and larger glucose excursions in the hour following meal intake(49). The dose of GLP-1 receptor antagonist (Exendin-(9-39) IV bolus of 7500 pmol/kg over 1 minute at Time 0 (Aim 1B) followed by continuous infusion of 750 pmol/kg/min for 150 minutes) was chosen as this dose elicits blockade of GLP-1 action at its receptor in healthy volunteers during a fixed blood glucose, as measured by augmented post-prandial glucagon secretion, a blunted increase in post-prandial insulin secretion, and a significant increase in post-prandial GLP-1 secretion.(40-42) The timing of Exendin-(9-39) infusion may be adjusted pending results of Aim1A to coincide with the timing of peak FBF response.
- 8. <u>L-N<sup>G</sup>-monomethyl arginine citrate (L-NMMA) (IND # \_\_\_\_\_\_)</u>- is an investigational agent (Clinalfa®, Bachem Distribution Services; Weil am Rhein, Germany) that will be infused intravenously. Side effects of systemic

administration include increase in blood pressure and decrease in heart rate. (3mg/kg priming IV infusion over 15 minutes given prior to Arginine infusion in Aim 1B and then continued at 6 mg/kg over an additional 120 minutes) has been selected to achieve peak hemodynamic response 15 minutes after priming dose and maintain hemodynamic effects for up to one hour after completion of infusion. (43;44)The elimination half-life of L-NMMA is approximately 60 minutes.(43) Co-infusion of a total dose of 6.5 mg/kg L-NMMA with L-arginine has not been shown to influence L-arginine stimulated GH secretion.(47) Doses up to 13.5 mg/kg IV have safely been given to healthy adults.(44-46)

# 7. Reporting of Adverse Events or Unanticipated Problems Involving Risk to Participants or Others

All adverse events and instances of non-compliance with the protocol, subject withdrawals, and subject complaints will be formally summarized and reviewed by the Data and Safety Monitoring Board (DSMB) bi- annually. The DSMB will receive these in written format and review the study for appropriate and timely subject accrual, adherence to the protocol, and data accuracy and completeness. The DSMB will provide the PI (Dr. Devin) with written confirmation of receipt of this bi-annual summary as well as a recommendation with accompanying rationale for study termination or continuation. This written confirmation will be provided to the IRB and include results of the review and concerns, if any, regarding subject safety or study drug tolerability. The DSMB will ensure that all adverse event reporting to the IRB is in

accordance with current policies. The members of the DSMB will be available for discussion of any questions regarding protocol adherence, consent issues, or adverse

events. The DSMB will review final results of the study.

The DSMB is comprised of Drs. is a translational researcher and has experience with the use of sitagliptin to treat patients with diabetes. Dr. is a translational researcher and has experience with the administration of vasoactive substances. All adverse events specifically related to the use of arginine and pegvisomant will be graciously reviewed as they occur with Dr., who as Director of Vanderbilt's Pituitary Center has extensive experience in the use of these agents to diagnose and treat patients with pituitary disease in the clinical setting. Dr. is a clinical endocrinologist and translational researcher at the University of Cincinnati who has experience with the infusion of exendin (9-39) in clinical research protocols. Dr. will serve as the DSMB chair.

is enrolled. Dr. Devin, her mentor (Dr. and her co-investigators will

closely oversee the protocol. Any serious adverse events or toxicities will be reported to the Vanderbilt IRB as per policy and will immediately be reviewed with the DSMB. Any noncompliance with the IRB-approved protocol that increases risk or affects participants' rights, safety or welfare will be reported to the IRB within 10 working days of the investigators' knowledge and immediately reviewed by the DSMB.

Any untoward medical event will be classified as an adverse event, regardless of its causal relationship with the study. An adverse event will be classified as serious if it a) results in death, b) if life-threatening, c) requires inpatient hospitalization or prolongation of existing hospitalization, d) results in persistent or significant disability or incapacity, e) is a congenital anomaly or birth defect. All non-serious adverse events and instances of non-compliance with the protocol will be reported annually to the IRB at the time of continuing review.

Dr. Devin will review enrollment progress, all adverse events, protocol adherence data, and data quality entry at a minimum of every two weeks with her mentor (Dr. Dr. Devin will review with Dr. each enrolled subject's chart every two weeks for side effects and tolerability of the investigational drug. These findings will be included in the DSMB bi-annual report unless dictated otherwise above.

Summary Reports will be submitted to the IRB at least annually and will contain a) the number of adverse events and an explanation of how each event was handled, b) the number of complaints and how each complaint was handled, c) the number of subject withdrawals and an explanation of why the subject withdrew or was withdrawn, and d) the number of protocol violations (non-compliance with protocol) and how each was handled.

### 8. Study Withdrawal/Discontinuation

If at any time during the study, a subject develops any symptoms related to study participation that subject will be withdrawn from the study. If, in the opinion of the investigator, a subject is non-compliant, that subject will be withdrawn from the study. Subjects who are withdrawn will be followed until symptoms have resolved.

### 9. Statistical Considerations

### Anticipated Results

DPPIV cleaves GRF at its penultimate alanine.(1;2) GRF stimulates endogenous GH secretion, potentially leading to an increase in the GH-mediated vasodilator response.(10;11) We expect that DPPIV inhibition (sitagliptin) will result in decreased degradation of GRF and an increase in stimulated GH secretion. (Aim 1A) We expect that this will increase forearm blood flow and that this effect will be prevented by pretreatment with a GH receptor antagonist, but remain unaffected by administration of L-NMMA as well as GLP-1 receptor antagonist. (Aim 1B)

### Sample Size and Power Calculation

Aim 1A. Our preliminary data in females (N=4) demonstrate a difference in mean peak GH following arginine stimulation of 6.79 ng/mL (mean 14.07 ± SD 4.73 ng/mL Drug A vs. 20.86 ± 13.23 ng/mL Drug B). Sample size was calculated with PS Software using the design for a paired t-test with a 0.05 two-sided significance level.(50) A sample size of 28 females will have 80% power to detect a difference in means of 6.79 ng/mL assuming a 12.25 ng/mL SD of the differences. Accounting for a 10% drop-out between the 2 study days, we will enroll 31 females in this study. Our preliminary data in males (N=2) demonstrates a difference in mean peak GH in the opposite direction. Premenopausal women are more responsive to GHRH and secrete more GH per pulse than men, the latter is primarily a GHRH-mediated phenomenon. (51-53) Given the known sexual dimorphism in pulsatile GH secretion, we have chosen to study only enough men to allow us to estimate the difference in males. Studying 11 males will allow a half-width of the 95% confidence for the difference to be about 7.6 ng/mL. Enrolling forty-four subjects (32 females; 12 males) in Aim 1A divided amongst 3 groups in Aim 1B will allow each group to be adequately powered to detect a statistically significant difference in FBF (see below).

Aim 1B. Prior data indicates that a difference in forearm blood flow of the following is statistically significant p<0.001: baseline forearm blood flow mean ±SEM 4.4 ±0.2 vs 2.7 ±0.3 ml/min/100mLfollowing L-NMMA in n=59 subjects. (54) Conservatively assuming a correlation coefficient of 0.6 for the two measures on the same subject, the SD for the within subject difference would be 1.8. Assuming, for example, that sitagliptin+GH antagonist would achieve FBF of 2.7 ± 2.3 and sitagliptin+placebo would have FBF of 4.4±1.5 (mean±SD), a sample size of 11 completed subjects would have 80% power to detect this difference. Sample size was calculated with PS Software using the design for a paired t-test. Assuming a 10% drop-out in between the 2 study visits we will enroll 14 patients in each Group; gender distribution of the groups will be determined by the results from Aim 1A.

### Data Analysis Plan

### The primary endpoints are:

**Aim 1A**: Peak GH level following Arginine stimulation, assessed in a paired manner with and without sitagliptin.

**Aim 1B**: Repeated measurements of FBF following sitagliptin at the specified times will be assessed in a paired manner with and without antagonist.

Even though we do not expect any carry-over effect in this 2 by 2 crossover study with repeated measures based upon our prior experience with studies of sitagliptin, we will first test for a carry-over effect using the T-test approach proposed by Jones and Kenward.(55) Mixed effect models will be used to analyze the data with a random subject effect and with the treatment (sitagliptin vs placebo or sitagliptin+GH antagonist vs sitagliptin+placebo) and the time trend as measured at the above time points as fixed effects. The focus of this study will be the treatment effect and the time trend of the endpoints; however, mixed effect models also provide the flexibility of controlling for and evaluating covariates as needed by the study. The mixed effect models are robust in the sense that they can include subjects with missing data at some time points but not all time points to estimate the effects of interest. The above specifies the general model for most of the endpoints, however, there will be no time trend in the model for peak GH level. Besides the above evaluation of the treatment effect and the time trend through the regression models, specific inferences regarding effects of interest will be made by reporting a point estimate along with a 95% confidence interval. Hypotheses will be tested at the level of  $\alpha$ =0.05. This data analysis plan will be carried out using statistical software SPSS for Windows (Version 19.0, SPSS, Chicago) and the open source statistical package R (version 2.12, R Development Core Team, 2006).

# 10. Privacy/Confidentiality Issues

Clinical data, including clinical laboratory, will be entered by a member of the Key Study Personnel in a protected source database (RedCap). A unique identification case number will be used to protect the confidentiality of the study participants. The case numbers and participants' names will be included in the protected source database, accessible only by Key Study Personnel, but only case numbers will be included in any spreadsheet used for the statistical analysis.

### 11. Follow-up and Record Retention

The total duration of enrollment will be 2 years, and we anticipate completion of a manuscript within 3 years of initiation. All records will be retained for 7 years following publication of the data. After that time, records may be archived for an additional 5 years and then shredded.

#### **Reference List**

- (1) Zhu L, Tamvakopoulos C, Xie D, Dragovic J, Shen X, Fenyk-Melody JE, et al. The role of dipeptidyl peptidase IV in the cleavage of glucagon family peptides: in vivo metabolism of pituitary adenylate cyclase activating polypeptide-(1-38). J Biol Chem 2003 Jun 20;278(25):22418-23.
- (2) Bongers J, Lambros T, Ahmad M, Heimer EP. Kinetics of dipeptidyl peptidase IV proteolysis of growth hormone-releasing factor and analogs. Biochim Biophys Acta 1992 Jul 31;1122(2):147-53.
- (3) Dzurik MV, Diedrich A, Black B, Paranjape SY, Raj SR, Byrne DW, et al. Endogenous substance P modulates human cardiovascular regulation at rest and during orthostatic load. J Appl Physiol 2007 Jun;102(6):2092-7.
- (4) Boerrigter G, Costello-Boerrigter LC, Harty GJ, Lapp H, Burnett JC, Jr. Des-serine-proline brain natriuretic peptide 3-32 in cardiorenal regulation. Am J Physiol Regul Integr Comp Physiol 2007 Feb;292(2):R897-R901.
- (5) Marney A, Kunchakarra S, Byrne L, Brown NJ. Interactive hemodynamic effects of dipeptidyl peptidase-IV inhibition and angiotensin-converting enzyme inhibition in humans. Hypertension 2010 Oct;56(4):728-33.
- (6) Mistry GC, Maes AL, Lasseter KC, Davies MJ, Gottesdiener KM, Wagner JA, et al. Effect of sitagliptin, a dipeptidyl peptidase-4 inhibitor, on blood pressure in nondiabetic patients with mild to moderate hypertension. J Clin Pharmacol 2008 May;48(5):592-8.
- (7) Shah Z, Pineda C, Kampfrath T, Maiseyeu A, Ying Z, Racoma I, et al. Acute DPP-4 inhibition modulates vascular tone through GLP-1 independent pathways. Vascul Pharmacol 2011 Jul;55(1-3):2-9.
- (8) Frohman LA, Downs TR, Heimer EP, Felix AM. Dipeptidylpeptidase IV and trypsin-like enzymatic degradation of human growth hormone-releasing hormone in plasma. J Clin Invest 1989 May;83(5):1533-40.
- (9) Vance ML. Growth-hormone-releasing hormone. Clin Chem 1990 Mar;36(3):415-20.

- (10) Napoli R, Guardasole V, Angelini V, D'Amico F, Zarra E, Matarazzo M, et al. Acute effects of growth hormone on vascular function in human subjects. J Clin Endocrinol Metab 2003 Jun;88(6):2817-20.
- (11) Li G, Del Rincon JP, Jahn LA, Wu Y, Gaylinn B, Thorner MO, et al. Growth hormone exerts acute vascular effects independent of systemic or muscle insulin-like growth factor I. J Clin Endocrinol Metab 2008 Apr;93(4):1379-85.
- (12) Schini-Kerth VB. Dual effects of insulin-like growth factor-I on the constitutive and inducible nitric oxide (NO) synthase-dependent formation of NO in vascular cells. J Endocrinol Invest 1999;22(5 Suppl):82-8.
- (13) Gornik HL, Creager MA. Arginine and endothelial and vascular health. J Nutr 2004 Oct;134(10 Suppl):2880S-7S.
- (14) Forstermann U, Sessa WC. Nitric oxide synthases: regulation and function. Eur Heart J 2011 Sep 1.
- (15) Thum T, Fleissner F, Klink I, Tsikas D, Jakob M, Bauersachs J, et al. Growth hormone treatment improves markers of systemic nitric oxide bioavailability via insulin-like growth factor-I. J Clin Endocrinol Metab 2007 Nov;92(11):4172-9.
- (16) Devin JK, Vaughan DE, Blevins LS, Jr., Chen Q, Covington J, Verity DK, et al. Low-dose growth hormone administration mobilizes endothelial progenitor cells in healthy adults. Growth Horm IGF Res 2008 Jun;18(3):253-63.
- (17) Thum T, Bauersachs J. Growth hormone regulates vascular function-what we know from bench and bedside. Eur J Clin Pharmacol 2006;62(Supplement 1):29-32.
- (18) Bulow B, Hagmar L, Mikoczy Z, Nordstrom CH, Erfurth EM. Increased cerebrovascular mortality in patients with hypopituitarism. Clin Endocrinol (Oxf) 1997 Jan;46(1):75-81.
- (19) Bulow B, Hagmar L, Eskilsson J, Erfurth EM. Hypopituitary females have a high incidence of cardiovascular morbidity and an increased prevalence of cardiovascular risk factors. J Clin Endocrinol Metab 2000 Feb;85(2):574-84.
- (20) Erfurth EM, Bulow B, Eskilsson J, Hagmar L. High incidence of cardiovascular disease and increased prevalence of cardiovascular risk factors in women with hypopituitarism not receiving growth hormone treatment: preliminary results. Growth Horm IGF Res 1999 Apr;9 Suppl A:21-4.
- (21) Devin JK, Blevins LS, Jr., Verity DK, Chen Q, Bloodworth JR, Jr., Covington J, et al. Markedly impaired fibrinolytic balance contributes to cardiovascular risk in adults with growth hormone deficiency. J Clin Endocrinol Metab 2007 Sep;92(9):3633-9.
- (22) Pfeifer M, Verhovec R, Zizek B, Prezelj J, Poredos P, Clayton RN. Growth hormone (GH) treatment reverses early atherosclerotic changes in GH-deficient adults. J Clin Endocrinol Metab 1999 Feb;84(2):453-7.

- (23) Colao A, Di SC, Pivonello R, Cuocolo A, Spinelli L, Bonaduce D, et al. The cardiovascular risk of adult GH deficiency (GHD) improved after GH replacement and worsened in untreated GHD: a 12-month prospective study. J Clin Endocrinol Metab 2002 Mar;87(3):1088-93.
- (24) Colao A, Di SC, Rota F, Pivonello R, Savanelli MC, Spiezia S, et al. Short-term effects of growth hormone (GH) treatment or deprivation on cardiovascular risk parameters and intima-media thickness at carotid arteries in patients with severe GH deficiency. J Clin Endocrinol Metab 2005 Apr;90(4):2056-62.
- (25) Weaver JU, Monson JP, Noonan K, John WG, Edwards A, Evans KA, et al. The effect of low dose recombinant human growth hormone replacement on regional fat distribution, insulin sensitivity, and cardiovascular risk factors in hypopituitary adults. J Clin Endocrinol Metab 1995 Jan;80(1):153-9.
- (26) Sesmilo G, Biller BM, Llevadot J, Hayden D, Hanson G, Rifai N, et al. Effects of growth hormone administration on inflammatory and other cardiovascular risk markers in men with growth hormone deficiency. A randomized, controlled clinical trial. Ann Intern Med 2000 Jul 18;133(2):111-22.
- (27) Smith JC, Evans LM, Wilkinson I, Goodfellow J, Cockcroft JR, Scanlon MF, et al. Effects of GH replacement on endothelial function and large-artery stiffness in GH-deficient adults: a randomized, double-blind, placebo-controlled study. Clin Endocrinol (Oxf) 2002 Apr;56(4):493-501.
- (28) Boger RH. Nitric oxide and the mediation of the hemodynamic effects of growth hormone in humans. J Endocrinol Invest 1999;22(5 Suppl):75-81.
- (29) Boger RH, Skamira C, Bode-Boger SM, Brabant G, von zur MA, Frolich JC. Nitric oxide may mediate the hemodynamic effects of recombinant growth hormone in patients with acquired growth hormone deficiency. A double-blind, placebo-controlled study. J Clin Invest 1996 Dec 15;98(12):2706-13.
- (30) Calver A, Collier J, Vallance P. Inhibition and stimulation of nitric oxide synthesis in the human forearm arterial bed of patients with insulin-dependent diabetes. J Clin Invest 1992 Dec;90(6):2548-54.
- (31) Toda N, Imamura T, Okamura T. Alteration of nitric oxide-mediated blood flow regulation in diabetes mellitus. Pharmacol Ther 2010 Sep;127(3):189-209.
- (32) Lam CS, Chen MH, Lacey SM, Yang Q, Sullivan LM, Xanthakis V, et al. Circulating insulin-like growth factor-1 and its binding protein-3: metabolic and genetic correlates in the community. Arterioscler Thromb Vasc Biol 2010 Jul;30(7):1479-84.
- (33) Cordido F, Garcia-Buela J, Sangiao-Alvarellos S, Martinez T, Vidal O. The decreased growth hormone response to growth hormone releasing hormone in obesity is associated to cardiometabolic risk factors. Mediators Inflamm 2010;2010:434562.

- (34) Devin JK, Pretorius M, Nian H, Yu C, Billings FT, Brown NJ. Substance P Increases Sympathetic Activity During Combined Angiotensin-Converting Enzyme and Dipeptidyl Peptidase-4 Inhibition. Hypertension 2014 Feb 10;63(5):951-7.
- (35) Baum HB, Biller BM, Katznelson L, Oppenheim DS, Clemmons DR, Cannistraro KB, et al. Assessment of growth hormone (GH) secretion in men with adult-onset GH deficiency compared with that in normal men--a clinical research center study. J Clin Endocrinol Metab 1996 Jan;81(1):84-92.
- (36) Biller BM, Samuels MH, Zagar A, Cook DM, Arafah BM, Bonert V, et al. Sensitivity and specificity of six tests for the diagnosis of adult GH deficiency. J Clin Endocrinol Metab 2002 May;87(5):2067-79.
- (37) Muller AF, Leebeek FW, Janssen JA, Lamberts SW, Hofland L, van der Lely AJ. Acute effect of pegvisomant on cardiovascular risk markers in healthy men: implications for the pathogenesis of atherosclerosis in GH deficiency. J Clin Endocrinol Metab 2001 Nov;86(11):5165-71.
- (38) Veldhuis JD, Bidlingmaier M, Anderson SM, Wu Z, Strasburger CJ. Lowering total plasma insulin-like growth factor I concentrations by way of a novel, potent, and selective growth hormone (GH) receptor antagonist, pegvisomant (B2036-peg), augments the amplitude of GH secretory bursts and elevates basal/nonpulsatile GH release in healthy women and men. J Clin Endocrinol Metab 2001 Jul;86(7):3304-10.
- (39) Muller AF, Janssen JA, Lamberts SW, Bidlingmaier M, Strasburger CJ, Hofland L, et al. Effects of fasting and pegvisomant on the GH-releasing hormone and GH-releasing peptide-6 stimulated growth hormone secretion. Clin Endocrinol (Oxf) 2001 Oct;55(4):461-7.
- (40) Salehi M, Prigeon RL, D'Alessio DA. Gastric bypass surgery enhances glucagon-like peptide 1-stimulated postprandial insulin secretion in humans. Diabetes 2011 Sep;60(9):2308-14.
- (41) Salehi M, Vahl TP, D'Alessio DA. Regulation of islet hormone release and gastric emptying by endogenous glucagon-like peptide 1 after glucose ingestion. J Clin Endocrinol Metab 2008 Dec;93(12):4909-16.
- (42) Salehi M, Aulinger B, Prigeon RL, D'Alessio DA. Effect of endogenous GLP-1 on insulin secretion in type 2 diabetes. Diabetes 2010 Jun;59(6):1330-7.
- (43) Mayer BX, Mensik C, Krishnaswami S, Derendorf H, Eichler HG, Schmetterer L, et al. Pharmacokinetic-pharmacodynamic profile of systemic nitric oxide-synthase inhibition with L-NMMA in humans. Br J Clin Pharmacol 1999 May;47(5):539-44.
- (44) Albert J, Schedin U, Lindqvist M, Melcher A, Hjemdahl P, Frostell C. Blockade of endogenous nitric oxide production results in moderate hypertension, reducing sympathetic activity and shortening bleeding time in healthy volunteers. Acta Anaesthesiol Scand 1997 Oct;41(9):1104-13.

- (45) Spahr L, Martin PY, Giostra E, Niederberger M, Lang U, Capponi A, et al. Acute effects of nitric oxide synthase inhibition on systemic, hepatic, and renal hemodynamics in patients with cirrhosis and ascites. J Investig Med 2002 Mar;50(2):116-24.
- (46) Hjorth LL, Klingenberg IH, Olesen J. A dose-response study of nitric oxide synthase inhibition in different vascular beds in man. Eur J Clin Pharmacol 2003 Oct;59(7):499-505.
- (47) Fisker S, Nielsen S, Ebdrup L, Bech JN, Christiansen JS, Pedersen EB, et al. L-arginine-induced growth hormone secretion is not influenced by co-infusion of the nitric oxide synthase inhibitor N-monomethyl-L-arginine in healthy men. Growth Horm IGF Res 1999 Feb;9(1):69-73.
- (48) Salehi M, Prigeon RL, D'Alessio DA. Gastric bypass surgery enhances glucagon-like peptide 1-stimulated postprandial insulin secretion in humans. Diabetes 2011 Sep;60(9):2308-14.
- (49) Deane AM, Nguyen NQ, Stevens JE, Fraser RJ, Holloway RH, Besanko LK, et al. Endogenous glucagon-like peptide-1 slows gastric emptying in healthy subjects, attenuating postprandial glycemia. J Clin Endocrinol Metab 2010 Jan;95(1):215-21.
- (50) Dupont WD, Plummer WD, Jr. Power and sample size calculations. A review and computer program. Control Clin Trials 1990 Apr;11(2):116-28.
- (51) Giustina A, Veldhuis JD. Pathophysiology of the neuroregulation of growth hormone secretion in experimental animals and the human. Endocr Rev 1998 Dec;19(6):717-97.
- (52) Goldenberg N, Barkan A. Factors regulating growth hormone secretion in humans. Endocrinol Metab Clin North Am 2007 Mar;36(1):37-55.
- (53) van den Berg G, Veldhuis JD, Frolich M, Roelfsema F. An amplitude-specific divergence in the pulsatile mode of growth hormone (GH) secretion underlies the gender difference in mean GH concentrations in men and premenopausal women. J Clin Endocrinol Metab 1996 Jul;81(7):2460-7.
- (54) Fong P, Stafforini DM, Brown NJ, Pretorius M. Increased blood flow induces oxidative stress through an endothelium- and nitric oxide-independent mechanism. Free Radic Biol Med 2010 Jul 15;49(2):301-5.
- (55) Jones B, Kenward MG. Design and Analysis of Crossover Trials. Boca Raton, FL: CRC Press LLC; 2003.